CLINICAL TRIAL: NCT05599737
Title: Stereotactic Prostate Radiotherapy With Dose Escalation Focused on the "Dominant Intra-prostatic Lesion" (DIPL) Delineated by Multi-parametric MRI and 68Ga-PSMA PET (Prostate-SIB-PSMA)
Acronym: Prostate-SIB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ET21-129
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-05

CONDITIONS: Prostate Adenocarcinoma
Keywords: Localized; Intermediate risk; Initial care; Not operated; Integrated boost; multiparametric MRI; Dominant Intra-Prostatic Lesion (DIPL); 68Ga-PSMA PET; Safety; Dosimetric planning; Recurrence
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiotherapy (Experimental): Stereotactic radiotherapy in 5 fractions (on alternate day)
  * Whole prostate: 36.25 Gy - 7.25Gy/fraction
  * GTV-RT (boost): target 50 Gy - 10 Gy/fraction
  Interventions: Radiation: Integrated boost

INTERVENTIONS:
Radiation: Integrated boost — Integrated boost based on the dominant intra-prostatic lesion delineated on multi-parametric Magnetic Resonance Imaging and 68Ga-Prostate Specific Membrane Antigen Positron Emission Tomography

SUMMARY:
In localized intermediate- and high-risk prostate cancers (according to the NCCN classification), external radiotherapy delivering a "high" dose (dose equivalent 78-80Gy EQD2, α/ß=1.5) to the entire prostate volume combined with hormonal treatment, if necessary, has shown its benefit in terms of recurrence-free survival and is considered a standard treatment for this indication.

Two fractionation modalities (number of sessions) are considered as therapeutic standards, conventional fractionation (39 to 40 sessions of 2 Gy in 8 weeks) and moderate hypo-fractionation (20 sessions of 3 Gy). More recently, phase II and two phase III studies have shown equivalence in terms of safety and efficacy of "extreme hypofractionation" (5 or 6 sessions) for these localized cancers, using stereotactic-type techniques. In view of the current data, this fractionation is considered a therapeutic standard in some countries (notably the USA) and an option in France.

Delivering higher doses, beyond 80 GyEQD2 would improve tumor control, as demonstrated by randomized studies using brachytherapy, but at the cost of an increased risk of urinary toxicity.

As an alternative to this combination of external radiotherapy and brachytherapy, an innovative approach of external radiotherapy has been developed to increase the therapeutic ratio of patients with localized prostate cancer, based on an escalation of the radiation dose (> 95 GyEQD2) focused on the macroscopic tumor or "dominant intra-prostatic lesion" (DIPL), the area most at risk of local recurrence after conventional dose radiotherapy (3). This external radiotherapy technique consists in performing a conventional dose irradiation on the whole prostate, with at the same time (at each session) a higher dose ("Boost") on the DIPL. This is a modality known as "simultaneous integrated boost" (SIB).

The feasibility of simultaneous integrated boost (SIB) on the DIPL has been proven in external radiotherapy using conventional fractionation in the phase III FLAME study and the results in terms of long-term tumor control of this study showed a benefit in terms of biological recurrence-free survival.

Feasibility in terms of tolerance has also been established for very hypofractionated regimens (5 sessions), in particular in the HypoFLAME study that followed the above-mentioned study .

Multiparametric MRI (mpMRI) is used to identify and delineate the "dominant intra-prostatic lesion" (DIPL), and is the most commonly used modality in clinical studies that have evaluated SIB techniques.

However, several studies show that PET imaging, particularly 68Ga-PSMA PET, significantly improves the correlation between the image-defined DIPL and histological data and may improve the likelihood of tumor control. A dosimetric simulation study also showed that dose escalation based on 68Ga-PSMA PET could improve local tumor control with an acceptable level of toxicity .

Moreover, 68Ga-PSMA PET could be used to select the patients who could benefit most from this dose escalation, by excluding patients with lymph node or distant metastases.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age is ≥ 18 years;
* Patient with intermediate-risk or high-risk prostate adenocarcinoma with a single severity criterion based on the NCCN classification
* Patient with at least 12 randomized biopsies
* N0 staging (CT or MRI or PET - choline) M0 (bone scan or PET - choline) with imaging workup less than 6 months old
* Dominant intra-prostate lesion identifiable on a recent multi-parametric MRI (< = 6 months) with an estimated volume < 40% of the entire prostate volume
* Informed patient who has signed a consent to participate in the study
* Patient enrolled in a health insurance plan (or beneficiary of such a plan)

Exclusion Criteria:

* Patient with pre-therapeutic micturition disorders (IPSS score > 15)
* Patient with digestive inflammatory disease
* Patient with high risk prostate adenocarcinoma with more than one severity criteria based on the NCCN classification
* Prostate volume > 60 cc
* Patient with hip replacement
* Patient with a contraindication to the implantation of fiduciary implants (anticoagulants that cannot be stopped for gold bead implantation)
* Patient with a contraindication to MRI
* Patient who has had a trans-urethral resection of the prostate within 3 months prior to inclusion
* History of previous pelvic radiotherapy
* Patient with previous hormonal treatment
* Known hypersensitivity to the active substance or to the excipients used for the 68Ga-PSMA PET
* Patient with a contraindication to the administration of Lasilix
* Patient for whom follow-up does not seem feasible even in the short term
* Patient participating in another clinical trial that may interfere with the evaluation of the primary endpoint
* Patient under guardianship or deprived of liberty.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-24 (Actual); Primary Completion 2024-05-25 (Estimated); Study Completion 2024-05-25 (Estimated)

PRIMARY OUTCOMES:
Tolerance of the treatment regimen | 12 Months
  Rate of patients with at least one acute toxicity ≥ grade 3 occurring up to 3 months post RT or one late toxicity ≥ grade 2 occurring from 3 months post RT according to the NCI-CTC-v5.0 scale and attributable to radiotherapy (Gastrointestinal or genitourinary toxicities)

SECONDARY OUTCOMES:
Change in the stage of the disease | 5-10 days after trustee implantation
  Proportion of patients excluded following 68Ga-PSMA PET (non-localised cancers or Index Tumour > 40% of prostate volume)
Dosimetric feasibility | During RT
  Dose delivered on DIPL and proportion of patients for whom dose escalation ≥ 95 GyEQD2 is possible
Adaptability of the 68Ga-PSMA PET preparation protocol to dosimetric planning | Before RT
  Confirmation that the 68Ga-PSMA PET preparation protocol is suitable for dosimetric planning
All grades toxicity | 12 Months
  Rate of all grades of toxicity according to NCI-CTC-v5.0
Tumour control | 12 Months
  Rate of patients with recurrence (biological, local or distant)

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Centre Marie Curie, Valence, Drôme
  - CAC-Clermont-Ferrand - Centre Jean Perrin, Clermont-Ferrand, Puy-de-Dôme
  - Hospices Civils de Lyon (Hôpital Edouard Herriot), Lyon, Rhône
  - Centre Léon Bérard, Lyon, Rhône